CLINICAL TRIAL: NCT00809211
Title: A Phase II Multi-center, Open-label, Study of Nilotinib at a Dose of 300mg Twice Daily in Adult Patients With Newly Diagnosed Philadelphia Chromosome Positive (Ph+) Chronic Myelogenous Leukemia in Chronic Phase (CML-CP)
Brief Title: Nilotinib in Treating Patients With Newly Diagnosed Chronic Phase Chronic Myelogenous Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Trials Ireland (Network)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICORG 08-02; ICORG 08-02; EUDRACT-2008-004551-30; EU-20899
Record Dates: First submitted 2008-12-16; First posted 2008-12-17 (Estimated); Last update posted 2018-07-24 (Actual); Status verified 2018-07

CONDITIONS: Leukemia
Keywords: chronic myelogenous leukemia, BCR-ABL1 positive; chronic phase chronic myelogenous leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Myeloid, Chronic-Phase | interventions — nilotinib; Cytogenetic Analysis; Polymerase Chain Reaction

ARMS (1):
- Nilotinib (Experimental)
  Interventions: Drug: nilotinib; Genetic: cytogenetic analysis; Genetic: mutation analysis; Genetic: polymerase chain reaction; Other: pharmacological study

INTERVENTIONS:
Drug: nilotinib
Genetic: cytogenetic analysis
Genetic: mutation analysis
Genetic: polymerase chain reaction
Other: pharmacological study

SUMMARY:
RATIONALE: Nilotinib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

PURPOSE: This phase II trial is studying how well nilotinib works in treating patients with newly diagnosed chronic phase chronic myelogenous leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To establish the complete cytogenetic response rate at 6 months in patients with newly diagnosed Philadelphia chromosome-positive chronic phase chronic myelogenous leukemia treated with nilotinib.

Secondary

* To establish the complete cytogenetic response rate at 3, 9, 12, 18, and 24 months in these patients.
* To establish the molecular response rate at 3, 6, 9, 12, 18, and 24 months in these patients.
* To establish the safety of this drug in these patients.
* To correlate pharmacokinetic data with response rate and toxicity.
* To correlate Bcr-Abl results using GeneXpert with Bcr-Abl results using international standardized quantitative PCR.
* To estimate the prevalence of Bcr-Abl mutations prior to and during treatment.

OUTLINE: This is a multicenter study.

Patients receive oral nilotinib twice daily on days 1-28. Treatment repeats every 28 days for up to 24 courses in the absence of disease progression or unacceptable toxicity.

Peripheral blood and bone marrow samples are collected periodically for mutation analysis, Bcr-Abl analysis by quantitative PCR, metaphase cytogenetics, and pharmacokinetic analysis.

After completion of study therapy, patients are followed every 3 months for 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Cytogenetically confirmed chronic myelogenous leukemia (CML) by standard conventional cytogenetic analysis of bone marrow*

  * Newly diagnosed disease (within the past 6 months) NOTE: *FISH cannot be used
* In chronic phase, as defined by the following:

  * Less than 15% blasts in peripheral blood and bone marrow
  * Less than 30% blasts plus promyelocytes in peripheral blood and bone marrow
  * Less than 20% basophils in peripheral blood
  * Platelet count ≥ 100,000/mm^3
  * No evidence of extramedullary leukemic involvement, except for hepatosplenomegaly
* Philadelphia chromosome-positive disease as demonstrated by (9;22) translocation (presence of Bcr-Abl)

  * A review of ≥ 20 metaphases is required
* No previously documented T315I mutations

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Total bilirubin < 1.5 times upper limit of normal (ULN)
* AST and ALT < 2.5 times ULN
* Estimated glomerular filtration rate ≥ 30 mL/min
* Serum amylase and lipase ≤ 1.5 times ULN
* Alkaline phosphatase ≤ 2.5 times ULN (unless related to CML)
* Potassium ≥ lower limit of normal (LLN)
* Magnesium ≥ LLN
* Phosphorous ≥ LLN
* Total calcium ≥ LLN (corrected for serum albumin)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No impaired cardiac function including, but not limited to, any of the following:

  * LVEF < 45% or < LLN by ECHO
  * Inability to determine the QT interval on ECG
  * Complete left bundle branch block
  * Congenital long QT syndrome or a known family history of long QT syndrome
  * History of or presence of clinically significant ventricular or atrial tachyarrhythmias
  * Clinically significant resting bradycardia (< 50 beats/min)
  * QTc > 450 msec on an average of 3 serial baseline ECGs (using the QTcF formula)
  * Clinically documented myocardial infraction within the past 12 months
  * Unstable angina within the past 12 months
  * Other clinically significant heart disease (e.g., congestive heart failure or uncontrolled hypertension)
* No severe or uncontrolled medical condition (e.g., uncontrolled diabetes or active or uncontrolled infection)
* No history of significant congenital or acquired bleeding disorder unrelated to CML
* No history of non-compliance to medical regimens
* No other primary malignancy unless it is neither currently clinically significant nor requiring active intervention
* No impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of the study drug (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, small bowel resection, or gastric bypass surgery)
* No acute pancreatitis within the past year
* No history of chronic pancreatitis
* No acute or chronic liver, pancreatic, or severe renal disease considered unrelated to CML

PRIOR CONCURRENT THERAPY:

* No prior therapy for CML other than hydroxyurea and/or anagrelide
* Prior imatinib mesylate allowed provided it was administered for ≤ 14 days
* More than 30 days since prior and no other concurrent investigational agents
* More than 4 weeks since prior major surgery and recovered
* No other concurrent anticancer agents, including chemotherapy and biologic agents
* No concurrent strong CYP3A4 inhibitors (e.g., erythromycin, ketoconazole, itraconazole, voriconazole, clarithromycin, telithromycin, ritonavir, mibefradil)
* No concurrent strong CYP3A4 inducers (e.g., dexamethasone, phenytoin, carbamazepine, rifampin, rifabutin, rifapentin, phenobarbital, St. John's wort)
* No concurrent medications that have the potential to prolong QT interval
* No concurrent grapefruit, star fruit, Seville oranges, or their derivatives

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2008-10; Primary Completion 2011-05 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Complete cytogenetic response rate at 6 months as assessed by metaphase analysis | 6 months

SECONDARY OUTCOMES:
Molecular response rate at 3, 6, 9, 12, 18, and 24 months as assessed by quantitative PCR | 6 months
Time to disease progression | 6 months
Duration of event-free survival | 6 months
Overall toxicity rate | 6 months
Correlation of pharmacokinetic data with response rate and toxicity | 6 months
Correlation of Bcr-Abl results using GeneXpert with Bcr-Abl results using international standardized quantitative PCR | 6 months
Prevalence of Bcr-Abl mutations prior to and during treatment | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Mike O'Dwyer, MD, Principal Investigator — University College London Hospitals
Locations (6):
- University of Texas Health Science Center at San Antonio, San Antonio, Texas, United States
- Universitätsklinikum Charité Berlin, Berlin, Germany
- Ireland (3):
  - Belfast City Hospital, Belfast
  - St. James's Hospital, Dublin
  - University College Hospital, Galway
- Chaim Sheba Medical Centre, Tel Litwinsky, Israel